CLINICAL TRIAL: NCT02456506
Title: Multiple Centre, Randomised, Controlled Trial of Hyperfractionated IMRT and Conventional Fraction IMRT for Patients With Loco-regionally Recurrent Nasopharyngeal Carcinoma.
Brief Title: Hyperfractionated Intensity-modulated Radiotherapy (IMRT) Versus Conventional Fraction IMRT for Patients With Loco-regionally Recurrent Nasopharyngeal Carcinoma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, MD, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU5010
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Nasopharyngeal Neoplasms; Mortality; Quality of Life; Complications
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperfractionated IMRT Group (Experimental): IMRT (total dose of 65Gy, division 54 times, twice a day, once 1.2Gy, irradiation interval of 6-8 hours)
  Interventions: Radiation: Hyperfractionated IMRT
- Conventional Fraction IMRT Group (Active Comparator): IMRT (total dose of 60Gy, division 27 times, once a day, every 2.2Gy)
  Interventions: Radiation: Conventional Fraction IMRT

INTERVENTIONS:
Radiation: Hyperfractionated IMRT
  Arms: Hyperfractionated IMRT Group
Radiation: Conventional Fraction IMRT
  Arms: Conventional Fraction IMRT Group

SUMMARY:
This study evaluates the hyperfractionated IMRT in the treatment of patients with locally recurrent nasopharyngeal carcinoma. Half of participants will receive hyperfractionated IMRT, while the other half will receive conventional fraction IMRT.

DETAILED DESCRIPTION:
Local recurrence is one of the most challenging issues faced with nasopharyngeal carcinoma (NPC) patients. 8.4% to 10.9% of the patients developed recurrent diseases at the primary or/and regional site after definitive radiotherapy. Although some patients with limited recurrent lesions underwent surgery, the main treatment for these recurrent NPC patients was still re-irradiation.

Multiple retrospective and prospective studies have reported: under the condition of conventional fraction IMRT with the total dose of 60 gray (Gy) (division 27 times, once a day, every 2.2Gy), you can get a better local tumor control rate and survival outcome. However, the patients still underwent some severe late complications including nasopharyngeal necrosis, nasopharyngeal bleeding, temporal lobe necrosis, with the incidence rates of 28.8%, 18.6%, 20.3%, respectively. Approximately 50% of recurrent NPC patients died of these severe late complications, significantly compromising the overall survival rate of the patients. Previous studies showed that hyperfractionated radiotherapy could reduce severe late complication rates significantly, without affecting the local control rate. Indeed, we found that under the condition of equal irradiation time and tumor equivalent dosage between hyperfractionated IMRT (total dose of 65Gy, division 54 times, twice a day, once 1.2Gy, irradiation interval of 6-8 hours) and conventional fraction IMRT (total dose of 60Gy, division 27 times, once a day, every 2.2Gy), the normal late responding tissues equivalent dosage( EQD2) significantly decreased compared with conventional fraction IMRT. Therefore, the use of hyperfractionated IMRT is expected to decrease severe late complications rates, thereby improving the quality of life and overall survival of patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically approved WHO III patients received radical radiotherapy initially before recurrence (irradiation dosage > 66 Gy).

the interval time between initial treatment and relapse more than 1 year. recurrent Tumor stage2-4(rT2-4) Node stage0-2(rN0-2) Metastasis stage0(rM0) (rT2-4N0-2M0), overall stage II-IVa according to 2009 American Joint Committee on Cancer (AJCC/UICC) Tumor, Node, and Metastasis (TNM) staging system.

a Karnofsky performance status (KPS) score more than 70.

Exclusion Criteria:

* a history of previous or synchronous malignant tumors. recurrent Node stage3(rN3), recurrent Metastasis stage1(rM1) according to 2009 AJCC/UICC TNM staging system.

positive surgical margin after neck dissection. patients suffered with severe mental illness. severe diseases of the lung and cardiovascular system. severe hepatic and renal dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2015-06; Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | 3 year
Severe late complications rate | 2 year

SECONDARY OUTCOMES:
Quality of life questionnaire | 2 year
Loco-regional relapse free survival rate | 3 year
Distant metastasis free survival rate | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University; Yi Pan, MD, PhD, Study Director — Guangdong Provincial People's Hospital; Dong-Ping Chen, MD, PhD, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Cummings BJ. Benefits of accelerated hyperfractionation for head and neck cancer. Acta Oncol. 1999;38(2):131-6. doi: 10.1080/028418699431528. PMID 10227432
- [Background] Jereczek-Fossa BA, Morra A, DeBraud F, Alterio D, Mazzetta C, Rocca A, Catalano G, Bianchi L, Pasetti M, Chiesa F, Bruschini R, Orecchia R. Hyperfractionated radiotherapy in locally advanced nasopharyngeal cancer. An analysis of 43 consecutive patients. Strahlenther Onkol. 2004 Jul;180(7):425-33. doi: 10.1007/s00066-004-1202-9. PMID 15241530
- [Background] Jian JJ, Cheng SH, Tsai SY, Yen KC, Chu NM, Chan KY, Tan TD, Cheng JC, Lin YC, Leu SY, Hsieh CI, Tsou MH, Lin CY, Huang AT. Improvement of local control of T3 and T4 nasopharyngeal carcinoma by hyperfractionated radiotherapy and concomitant chemotherapy. Int J Radiat Oncol Biol Phys. 2002 Jun 1;53(2):344-52. doi: 10.1016/s0360-3016(02)02709-8. PMID 12023138
- [Background] Toita T, Ogawa K, Kamata M, Kojya S, Itokazu T, Kakinohana Y, Iraha S, Yoshinaga M, Zukeran Y, Sawada S. Hyperfractionated radiotherapy followed by adjuvant chemotherapy for nasopharyngeal cancer: report of seven cases. Jpn J Clin Oncol. 1999 Mar;29(3):160-3. doi: 10.1093/jjco/29.3.160. PMID 10225700
- [Derived] You R, Liu YP, Xie YL, Lin C, Duan CY, Chen DP, Pan Y, Qi B, Zou X, Guo L, Cao JY, Zhang YN, Wang ZQ, Liu YL, Ouyang YF, Wen K, Yang Q, Xie RQ, Li HF, Duan XT, Ding X, Peng L, Chen SY, Liang JL, Feng ZK, Xia TL, Xie RL, Jiang R, Gu CM, Liu RZ, Sun R, Yang X, Liu LZ, Ling L, Liu Q, Ng WT, Hua YJ, Huang PY, Chen MY. Hyperfractionation compared with standard fractionation in intensity-modulated radiotherapy for patients with locally advanced recurrent nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2023 Mar 18;401(10380):917-927. doi: 10.1016/S0140-6736(23)00269-6. Epub 2023 Feb 23. PMID 36842439